CLINICAL TRIAL: NCT01858675
Title: Predictive Value of Biomarkers on Volemia, Extra and Intra Vascular Varation and Hydroelectrolytic Disorders in Different ICU Patients
Brief Title: Biomarkers Correlation With Volemia
Acronym: ENVOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThermoFisher Scientific Brahms Biomarkers France (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A01310-41
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Cerebral Hemorrhage; Head Injury; Non Traumatic Post Surgery; Poly Trauma Patients Without Heart Failure; Renal Insufficiency
Keywords: ProADM; ProANP; proendothelin; proAVP; Cr 51; Volemia; fluid management; ICU patients; poly trauma patients
MeSH Terms: conditions — Cerebral Hemorrhage; Craniocerebral Trauma; Renal Insufficiency | interventions — Biomarkers; Erythrocyte Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biomarkers, total blood volume (Experimental)
  Interventions: Other: Biomarkers, red blood cells and plasma assessment

INTERVENTIONS:
Other: Biomarkers, red blood cells and plasma assessment

SUMMARY:
The purpose of this study is to determine whether the Biomarkers (pro adrenomedullin (MR proADM), pro arginin vasopressin (CT proAVP), pro atrial natriuretic peptid (MR proANP), Pro Endothelin) changes at Day 2, Day 5 and Day 7 of ICU admission are correlated with Intravascular volume assessed by Cr 51 on red blood cells (Day 2 and Day 7) and by I 125 on albumine Day 7. The correlation of these Biomarkers are also evaluted with other markers such as erythropoietin and catecholamines. 80 ICU patients are included.

ELIGIBILITY:
Inclusion Criteria:

* 20 Cerebral Hemorrhage
* 20 Head Injury
* 20 post surgery non traumatic non neuro
* 20 Polytrauma patients

Exclusion Criteria:

* Heart failure NYHA III or IV
* Renal insufficiency creatinin clearance < 30 ml/mn
* age < 18 Y
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Predictive value of biomarkers changes in Volemia variation | at Day 2, Day 5 and Day 7 of ICU admission
  Correlation with total blood volume(assessed by Cr 51) and biomarkers(Mr proADM, Mr proANP, CT proAVP and proendothelin)changes

SECONDARY OUTCOMES:
Predictive value of biomarkers changes with efficient volemia, fluid managements and other Markers such erythropoietin | at Day 2, Day 5 and Day 7 of ICU admission
  Correlation with efficient volemia and Biomarkers ( Mr proADM, Mr proANP, CT proAVP and proendothelin)changes.
Predictive value of Biomarkers with APACHE II and SOFA score and Prognosis at ICU discharge | at Day 2 , Day 5 and Day 7 of ICU admission and at discharge
  Correlation of Biomarkers changes with APACHE II and SOFA score and Mortality at Day 2, Day 5 and Day 7 of their ICU admission and at ICU discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Bicêtre, Le Krémilin Bicêtre, Île-de-France Region, France

REFERENCES:
- [Derived] Vigue B, Leblanc PE, Moati F, Pussard E, Foufa H, Rodrigues A, Figueiredo S, Harrois A, Mazoit JX, Rafi H, Duranteau J. Mid-regional pro-adrenomedullin (MR-proADM), a marker of positive fluid balance in critically ill patients: results of the ENVOL study. Crit Care. 2016 Nov 9;20(1):363. doi: 10.1186/s13054-016-1540-x. PMID 27825364